CLINICAL TRIAL: NCT04781400
Title: Bidirectional, Upbeat Communication and Differentiated, Distanced Care for Young People
Acronym: BUDDY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Desmond Tutu HIV Foundation (Other)
Collaborators: ViiV Healthcare (Industry); Karolinska Institutet (Other); University of North Carolina, Chapel Hill (Other); University of KwaZulu (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 448/2020
Record Dates: First submitted 2021-02-22; First posted 2021-03-04 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: HIV Infections; Covid19; Health Care Utilization; Gender-based Violence
MeSH Terms: conditions — HIV Infections; COVID-19; Patient Acceptance of Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote service delivery model PLUS mobile phone support (Experimental): Remote service delivery plus mobile intervention via SMS will include weekly check-ins from study staff, calls from a trained counsellor on request, and access to a two-way messaging feature.
  Interventions: Behavioral: Mobile phone support; Behavioral: Remote service delivery model
- Remote service delivery model (Active Comparator): Remote service delivery model.
  Interventions: Behavioral: Remote service delivery model

INTERVENTIONS:
Behavioral: Mobile phone support — Mobile phone support (SMS)
  Arms: Remote service delivery model PLUS mobile phone support
Behavioral: Remote service delivery model — ART treatment delivery via a courier service

SUMMARY:
Sub Saharan Africa is home to only 12% of the population, but accounts for approximately 70% of the global burden of HIV infection and 84% of infections among young people aged 10-24 years. South Africa, which currently has the largest SARS-CoV-2 pandemic in SSA, also has the largest HIV epidemic globally. Access and service delivery barriers to engaging in HIV care have contributed to estimates that only 49% of adolescents (aged 10-19 years) entering care from 2005-2016 have initiated antiretroviral therapy (ART). In response to the SARS-CoV-2 pandemic the South African government has implemented national lock-down orders that we predict will further inhibit treatment engagement among young people. Research is needed to identify best practices for safely retaining young people living with HIV (YPLWH) in care during COVID-19.

DETAILED DESCRIPTION:
The primary objectives of this study are to examine the feasibility, acceptability, and preliminary efficacy of a remote service delivery model for young people living with HIV aged 13-24 years that will include a monthly service needs assessment and optional delivery of HIV treatment services. YPLWH will also be randomized to receive (or not receive) mobile check-ins from study staff and access to two-way messaging capabilities to obtain continuous support for adherence to ART and COVID-19 prevention guidelines.

Investigators will also assess the impact of the COVID-19 lock-down orders on multi-level factors (individual, socio-behavioral, structural) over time among young people aged 13-24 years living with HIV (same cohort as above) and without HIV. Particular focus will be given to experience and perpetration of gender based violence. In addition, investigators will assess the impact of multi-level factors on compliance with COVID-19 prevention guidelines, health service utilization, and engagement in HIV care (YPLWH only). Findings will be examined overall and stratified by HIV status and gender.

Ultimately investigators hope to: (i) determine whether a remote service delivery model will help retain young people in HIV care and (ii) Inform the development of an intervention for young people in the study communities who may be experiencing GBV and associated outcomes in the wake of the pandemic.

ELIGIBILITY:
Inclusion Criteria:

Young people living with HIV who meet all of the following criteria will be eligible for inclusion into this study:

1. Speak isiXhosa and or English, residing in the Khayelitsha /Mitchell's Plain area
2. 13-24 years (inclusive)
3. Willing and able to provide informed telephonic or in person consent
4. Initiated ART at one of two health facilities and are currently in HIV care (i.e. received ART and had a viral load measurement in the past six months)
5. Regular access to a mobile phone with SMS or WhatsApp capacity (can include the phone of a parent/caregiver if the participant is <18 years or does not have their own phone)

Young people living without HIV from the same communities who meet all of the following criteria will be eligible for inclusion into this study:

1. Speak isiXhosa and or English, residing in the Khayelitsha / Mitchell's Plain area
2. 13-24 years (inclusive)
3. Willing and able to provide informed telephonic or in person consent
4. Has not previously tested positive for HIV and self-reports being HIV negative (i.e., not known to be living with HIV).
5. Regular access to a mobile phone (can include the phone of a parent/caregiver if the participant is <18 years or does not have their own phone)

Exclusion Criteria:

Young people living with HIV who meet any of the following criteria will be excluded from this study:

1. Not 13-24 years (inclusive)
2. Unwilling or unable to provide informed telephonic or in person consent
3. Not currently receiving ART care at a Desmond Tutu Health Foundation health facility
4. No regular access to a mobile phone with SMS or WhatsApp capacity
5. Planning to relocate in the next 6 months

Young people living without HIV from the same communities who meet any of the following criteria will be excluded this study:

1. Not 13-24 years (inclusive)
2. Unwilling or unable to provide informed telephonic or in person consent
3. Previously tested positive for HIV or is known to be living with HIV
4. No regular access to a mobile phone
5. Planning to relocate in the next 6 months

Ages: 13 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 536 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2022-05-13 (Actual); Study Completion 2022-05-13 (Actual)

PRIMARY OUTCOMES:
Acceptability of a remote service delivery and mobile support intervention assessed by the number of participants opting in to receive courier delivery of ART. | 6 months
  Program evaluation of a remote service delivery including mobile support intervention and courier delivery of ART amongst young people living with HIV.
Engagement in HIV care assessed by serial measurements of HIV Viral load. | 6 months
  Measurement of HIV viral load will be done at baseline, month three and month six to determine whether adherence to ART has been met (decrease or increase in HIV Viral load)
Changes in Gender Based Violence (GBV) incidence as a result of COVID lock-down measures as assessed by self reported surveys. | 6 months
  Investigate changes in self-reported GBV experience or perpetration, and other individual, social-behavioral, and structural factors that have been impacted by COVID-19 lock down orders.

SECONDARY OUTCOMES:
Incidence of COVID-19 infection by assessing participant IgG antibody levels. | 6 months
  Retrospective COVID-19 antibody testing at baseline and month
Qualitative themes assessed from in-depth individual interview data | 6 months
  Qualitative interviews will be used to inform intervention utility and the development of an intervention to reduce GBV

CONTACTS AND LOCATIONS:
Overall Officials: Linda-Gail Bekker, Principal Investigator — Desmond Tutu HIV Foundation
Locations (1):
- Gugulethu Community Health Centre, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: No